CLINICAL TRIAL: NCT02304861
Title: Viscoat Versus Visthesia. A Comparative Study of Post-cataract Endothelial Cell Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Democritus University of Thrace (Other)
Responsible Party: Principal Investigator, Georgios Labiris, Assistant Professor, Democritus University of Thrace
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: visco07012eit
Record Dates: First submitted 2014-11-11; First posted 2014-12-02 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Cataract
Keywords: cataract; viscoelastic (OVD) technology; endothelial cell count; endothelial cell pattern; central corneal edema
MeSH Terms: conditions — Cataract | interventions — chondroitin sulfate, sodium hyaluronate drug combination; visthesia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Viscoat group (Active Comparator): Patients operated using Viscoat OVD
  Interventions: Procedure: Viscoat
- Visthesia group (Active Comparator): Patients operated using Visthesia OVD
  Interventions: Procedure: Visthesia

INTERVENTIONS:
Procedure: Viscoat — Cataract extraction surgery performed with the Alcon Infiniti VisionSystem platform. Pupils were dilated with Tropicamide 0.5% (Tropixal, Demo, Greece) and Phenylephrine Hydrochloride 5% (Phenylephrine, Cooper, Greece). Periorbital skin and the lids were cleaned and the conjuctival cul-de-sac was irrigated with povidone iodine (Betadine). Patients received topical anesthesia with propacaine hydrochloride 0.5% drops (3 drops prior to surgery). By means of a 2.75mm, superior-temporal (eleven o'clock), self-sealing, clear-cornea incision 3% Sodium Hyaluronate, 4% Chondroitin Sulfate (Viscoat, Alcon, Greece) was injected in the anterior chamber
  Arms: Viscoat group
Procedure: Visthesia — Cataract extraction surgery performed with the Alcon Infiniti VisionSystem platform. Pupils were dilated with Tropicamide 0.5% (Tropixal, Demo, Greece) and Phenylephrine Hydrochloride 5% (Phenylephrine, Cooper, Greece). Periorbital skin and the lids were cleaned and the conjuctival cul-de-sac was irrigated with povidone iodine (Betadine). Patients received topical anesthesia with propacaine hydrochloride 0.5% drops (3 drops prior to surgery). By means of a 2.75mm, superior-temporal (eleven o'clock), self-sealing, clear-cornea incision sodium hyaluronate 1.5% and lidocaine hydrochloride 1% ophthalmic viscosurgical device (OVD) (Visthesia, Carl Zeiss, Germany) was injected in the anterior chamber
  Arms: Visthesia group

SUMMARY:
Objective of this study is the comparative assessment of the beneficial impact of the Viscoat viscoelastic (OVD) and Visthesia OVD on endothelial cells and corneal edema following torsional-ip cataract extraction surgery.

Participants will be recruited from the Cataract Service of the University Hospital of Alexandroupolis (UHA) in a consecutive-if-eligible basis. Eligibility criteria include diagnosis of senile cataract with stage 3 nuclear opalescence according to the Lens Opacities Classification System III (LOCS-3) grading scale. By means of a custom computer randomization program all participants will randomly populate two study groups according to the OVD used (ie. viscoat or visthesia).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of senile cataract with stage 3 nuclear opalescence according to the - Lens Opacities Classification System III (LOCS-3) grading scale

Exclusion Criteria:

* Endothelial cell count less than 1900,
* glaucoma,
* IOP-lowering medications,
* former incisional surgery,
* former diagnosis of corneal disease,
* diabetes or autoimmune diseases

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-01; Primary Completion 2014-06 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Endothelial Cell Count (ECD) | 3 months postoperatively

SECONDARY OUTCOMES:
Endothelial Cell pattern (ECP) | 3 months postoperatively
Central corneal edema (CCE) | 3 months postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Georgios Labiris, MD, PhD, Principal Investigator — Democritus University of Thrace
Locations (1):
- University Hospital of Alexandroupolis, Alexandroupoli, Evros, Greece

REFERENCES:
- [Result] Labiris G, Sideroudi H, Rousopoulos K, Kozobolis VP. Cohesive versus dispersive-cohesive ophthalmic viscosurgical device in torsional intelligent phaco. J Cataract Refract Surg. 2015 Mar;41(3):681-2. doi: 10.1016/j.jcrs.2015.01.010. No abstract available. PMID 25804586